CLINICAL TRIAL: NCT07192328
Title: Randomized Cross-Over Dose-Efficacy Study of rTMS in Healthy Young Female Volunteers
Brief Title: Dose-Efficacy of rTMS in Healthy Young Female Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Mataró (Other)
Responsible Party: Principal Investigator, Lluís Mundet, Principal Investigator GI Motility Unit, Hospital de Mataró
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IF04-03/2021; PERIS grant (SLT017/20/000125) (Other Grant/Funding Number: Departament de Salut de la Generalitat de Catalunya); PERIS grant SLT017/20/000236 (Other Grant/Funding Number: Departament de Salut de la Generalitat de Catalunya); ICI (ICI20/00117) (Other Grant/Funding Number: Instituto de Salud Carlos III, Barcelona, Spain)
Record Dates: First submitted 2025-09-16; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Fecal Incontinence (FI); Healthy Female Volunteer
Keywords: Motor Evoked Potentials; Healthy Volunteers; Neuromodulation; Transcranial Magnetic Stimulation; Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence | interventions — Transcranial Magnetic Stimulation; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: This was a randomized cross-over dose-response study conducted at the GI Motility Unit, Hospital de Mataró (Barcelona, Spain), in healthy young female volunteers aged 18-35 years. Exclusion criteria included pregnancy or potential for pregnancy, presence of a pacemaker, history of epilepsy or neurosurgery, study withdrawal, and poor treatment tolerance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- rTMS 1Hz (Experimental): rTMS delivered with 250 pulses via double-cone coil at either 1 Hz
  Interventions: Device: rTMS and rTLSMS administered using a Magstim Rapid2 repetitive stimulator at pre-identified hotspots (cortical, lumbar, and sacral regions bilaterally).
- rTMS 5Hz (Experimental): rTMS delivered with 250 pulses via double-cone coil at either 5 Hz
  Interventions: Device: rTMS and rTLSMS administered using a Magstim Rapid2 repetitive stimulator at pre-identified hotspots (cortical, lumbar, and sacral regions bilaterally).
- rTLSMS 1Hz (Experimental): rTLSMS (lumbar and sacral), 2400 pulses (600 per hotspot) applied at 1 Hz, using a 70mm refrigerated air film coil
  Interventions: Device: rTMS and rTLSMS administered using a Magstim Rapid2 repetitive stimulator at pre-identified hotspots (cortical, lumbar, and sacral regions bilaterally).
- rTLSMS 5Hz (Experimental): rTLSMS (lumbar and sacral), 2400 pulses (600 per hotspot) applied at 5 Hz, using a 70mm refrigerated air film coil
  Interventions: Device: rTMS and rTLSMS administered using a Magstim Rapid2 repetitive stimulator at pre-identified hotspots (cortical, lumbar, and sacral regions bilaterally).
- rTLSMS 10Hz (Experimental): rTLSMS (lumbar and sacral), 2400 pulses (600 per hotspot) applied at 10 Hz, using a 70mm refrigerated air film coil
  Interventions: Device: rTMS and rTLSMS administered using a Magstim Rapid2 repetitive stimulator at pre-identified hotspots (cortical, lumbar, and sacral regions bilaterally).

INTERVENTIONS:
Device: rTMS and rTLSMS administered using a Magstim Rapid2 repetitive stimulator at pre-identified hotspots (cortical, lumbar, and sacral regions bilaterally). — rTMS and rTLSMS administered using a Magstim Rapid2 repetitive stimulator at pre-identified hotspots (cortical, lumbar, and sacral regions bilaterally. rTMS delivered with 250 pulses via the same double-cone coil used for the neurophysiological study, at either 1 Hz or 5 Hz. For rTLSMS (lumbar and sacral), 2400 pulses (600 per hotspot) were applied at 1 Hz, 5 Hz, or 10 Hz using a 70mm refrigerated air film coil (Magstim, UK). Each dose and stimulation site (cortical or peripheral) were tested in separate sessions.
  Other Names: rTMS; Neurostimulation; Neuromodulation

SUMMARY:
This study is aimed to develop a new therapy based on non-invasive repetitive magnetic stimulation rehabilitation for FI in patients who do not respond to conventional therapies.

DETAILED DESCRIPTION:
AIMS 1) General: to develop a new therapy based on non-invasive repetitive magnetic stimulation rehabilitation for FI in patients who do not respond to conventional therapies. 2) Specific: a) To evaluate the optimal dose of cortical magnetic stimulation (rTMS) and lumbosacral magnetic stimulation (rTLS) in young healthy women for its subsequent application in patients with FI. b) To assess the effect of rTMS and rTLS on continence, clinical severity, and QoL in women with FI.

DESIGN: 1. Cross-over clinical trial dose-efficacy study: Evaluation of the dose-efficacy of acute rTMS and rTLS in 30 healthy young women. Frequencies will be evaluated for cortical rTMS (1Hz and 5Hz) and 3 rTLS (1, 5, and 10Hz).

ELIGIBILITY:
Inclusion Criteria:

* no history of FI
* Be a woman
* capable of understanding and providing informed consent

Exclusion Criteria:

* pregnancy and the ability to become pregnant
* presence of a pacemaker
* history of epilepsy or neurosurgery
* poor treatment tolerance

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
MEP Latency | Baseline (immediately before stimulation) and immediately after stimulation in each session, across 5 weekly sessions (up to 5 weeks).
  Latency from the onset of the stimuli (cortical or lumbosacral) to the first deflection of the MEP waveform.

SECONDARY OUTCOMES:
MEP amplitude | Baseline (immediately before stimulation) and immediately after stimulation in each session, across 5 weekly sessions (up to 5 weeks).
  Amplitude measured peak-to-peak of the MEP waveform.

CONTACTS AND LOCATIONS:
Overall Officials: Lluís Mundet, RN, PhD, Principal Investigator — Hospital de Mataró; Pere Clavé, MD, PhD, Principal Investigator — Hospital de Mataró
Locations (1):
- Hospital de Mataró, Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Sharing individual participant data is a decision we still have not taken

REFERENCES:
- [Background] Rao SSC, Yan Y, Xiang X, Sharma A, Ayyala D, Hamdy S. Effects of Translumbosacral Neuromodulation Therapy on Gut and Brain Interactions and Anorectal Neuropathy in Fecal Incontinence: A Randomized Study. Neuromodulation. 2021 Oct;24(7):1269-1277. doi: 10.1111/ner.13485. Epub 2021 Jun 22. PMID 34156730
- [Background] Tantiphlachiva K, Attaluri A, Valestin J, Yamada T, Rao SS. Translumbar and transsacral motor-evoked potentials: a novel test for spino-anorectal neuropathy in spinal cord injury. Am J Gastroenterol. 2011 May;106(5):907-14. doi: 10.1038/ajg.2010.478. Epub 2011 Jan 25. PMID 21266960
- [Background] Xiang X, Patcharatrakul T, Sharma A, Parr R, Hamdy S, Rao SSC. Cortico-anorectal, Spino-anorectal, and Cortico-spinal Nerve Conduction and Locus of Neuronal Injury in Patients With Fecal Incontinence. Clin Gastroenterol Hepatol. 2019 May;17(6):1130-1137.e2. doi: 10.1016/j.cgh.2018.09.007. Epub 2018 Sep 10. PMID 30213585